CLINICAL TRIAL: NCT06803225
Title: ULTRASOUND ASSESSMENT of GASTRIC CONTENT in FASTED PREGNANT WOMEN: PROSPECTIVE OBSERVATIONAL STUDY
Brief Title: Ultrasound Assessment of Gastric Volume in High-Risk Pregnant Women At Term
Status: Not yet recruiting | Type: Observational
Sponsor: The Chaim Sheba Medical Center (Other)
Responsible Party: Principal Investigator, Maxim Glebov, Dr., The Chaim Sheba Medical Center
Other Study IDs: 1346-24-SMC
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy; Respiratory Aspiration of Gastric Content

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Two-dimensional portable ultrasound unit with a low frequency (2-5 MHz) curved array transducer — Two-dimensional portable ultrasound unit with a low frequency (2-5 MHz) curved array transducer

SUMMARY:
The risk of pulmonary aspiration of gastric contents remains a significant risk during anesthesia, especially in pregnant women, as they may often require surgery without having observed appropriate fasting. A bedside ultrasound assessment of the status of the gastric content would be of great value for the clinician.

This prospective observational study aimed to (1) qualitatively and quantitatively describe the sonographic appearance of the gastric antrum in fasted high-risk pregnant women during the third trimester and (2) evaluate the relationship between demographic and clinical variables and the gastric antral cross-sectional area (CSA).

DETAILED DESCRIPTION:
The aim of this prospective study is to provide a qualitative and quantitative description of the sonographic appearance of the gastric antrum in fasted high-risk pregnant women in the 3rd trimester.

The investigators expect that the information obtained from the systematic ultrasonographic qualitative/quantitative assessment of the gastric content may help anesthesiologist to better assess aspiration risk and guide anesthetic and airway management, particularly in pregnant women scheduled for elective Cesarean delivery after standard preoperative fasting guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Non-labouring pregnant women at 3rd trimester (≥ 28 weeks)
2. 18 years or older.
3. ASA physical status I-III
4. Hospitilized in High Risk Pregnancy Department
5. Ability to understand the rationale of the study assessments and provide signed informed consent.
6. Written informed consent

Exclusion Criteria:

1. Patients with American Society of Anesthesiology (ASA) physical status class IV.
2. Patient age < 18 years
3. Pregnant patients with upper gastrointestinal (GI) disease and pathology.
4. History of upper GI tract surgical procedures.
5. History of medications that affect gastrointestinal motility.
6. Inability to understand the rationale of the study assessments and provide signed informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fasted (6h solids, 2h fluids) high-risk pregnant women at 3rd trimester
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative assessment of the antrum of the stomach | 10 min
  Patients will be classified as follows; Grade 0: the antrum appears empty on both supine and right lateral decubitus positions; grade 1: gastric fluid is visible on the right lateral decubitus position only, suggesting a small fluid volume; and grade 2: gastric fluid is observed in the antrum in both supine and right lateral decubitus, suggesting a larger fluid volume.

SECONDARY OUTCOMES:
Quantitative assessment of the antrum of the stomach | 10 min
  Three consecutive measures of the CSA (cross sectional area) of the antrum will be calculated via the ultrasound machine (free tracing method).

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data due to a specific request from our institution, which prioritises maintaining the confidentiality and privacy of patient information. The hospital's data-sharing policies and regulatory constraints are designed to safeguard sensitive health data and prevent potential risks of participant re-identification, even after anonymisation.

REFERENCES:
- [Background] Practice Guidelines for Obstetric Anesthesia: An Updated Report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia and the Society for Obstetric Anesthesia and Perinatology. Anesthesiology. 2016 Feb;124(2):270-300. doi: 10.1097/ALN.0000000000000935. No abstract available. PMID 26580836
- [Background] Perlas A, Arzola C, Van de Putte P. Point-of-care gastric ultrasound and aspiration risk assessment: a narrative review. Can J Anaesth. 2018 Apr;65(4):437-448. doi: 10.1007/s12630-017-1031-9. Epub 2017 Dec 11. PMID 29230709
- [Background] Roukhomovsky M, Zieleskiewicz L, Diaz A, Guibaud L, Chaumoitre K, Desgranges FP, Leone M, Chassard D, Bouvet L; AzuRea, CAR'Echo Collaborative Networks. Ultrasound examination of the antrum to predict gastric content volume in the third trimester of pregnancy as assessed by MRI: A prospective cohort study. Eur J Anaesthesiol. 2018 May;35(5):379-389. doi: 10.1097/EJA.0000000000000749. PMID 29210844
- [Background] Zieleskiewicz L, Bouvet L, Einav S, Duclos G, Leone M. Diagnostic point-of-care ultrasound: applications in obstetric anaesthetic management. Anaesthesia. 2018 Oct;73(10):1265-1279. doi: 10.1111/anae.14354. Epub 2018 Jul 26. PMID 30047997
- [Background] Kruisselbrink R, Gharapetian A, Chaparro LE, Ami N, Richler D, Chan VWS, Perlas A. Diagnostic Accuracy of Point-of-Care Gastric Ultrasound. Anesth Analg. 2019 Jan;128(1):89-95. doi: 10.1213/ANE.0000000000003372. PMID 29624530
- [Background] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Background] Dean G, Jacobs AR, Goldstein RC, Gevirtz CM, Paul ME. The safety of deep sedation without intubation for abortion in the outpatient setting. J Clin Anesth. 2011 Sep;23(6):437-42. doi: 10.1016/j.jclinane.2011.05.001. Epub 2011 Aug 9. PMID 21831622
- [Background] D'Angelo R, Smiley RM, Riley ET, Segal S. Serious complications related to obstetric anesthesia: the serious complication repository project of the Society for Obstetric Anesthesia and Perinatology. Anesthesiology. 2014 Jun;120(6):1505-12. doi: 10.1097/ALN.0000000000000253. PMID 24845921
- [Background] Neelakanta G, Chikyarappa A. A review of patients with pulmonary aspiration of gastric contents during anesthesia reported to the Departmental Quality Assurance Committee. J Clin Anesth. 2006 Mar;18(2):102-7. doi: 10.1016/j.jclinane.2005.07.002. PMID 16563326
- [Background] MENDELSON CL. The aspiration of stomach contents into the lungs during obstetric anesthesia. Am J Obstet Gynecol. 1946 Aug;52:191-205. doi: 10.1016/s0002-9378(16)39829-5. No abstract available. PMID 20993766